CLINICAL TRIAL: NCT05222997
Title: Therapy of Age-related Macular Degeneration Through Training With the Medical Eye Trainer
Brief Title: Therapy of Age-related Macular Degeneration
Acronym: MET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Robert Hörantner (Other)
Responsible Party: Sponsor-Investigator, Robert Hörantner, Head of Ophthalmology, Krankenhaus der Barmherzigen Schwestern Ried
Organization: Krankenhaus der Barmherzigen Schwestern Ried (Other)
Other Study IDs: 1241/2021
Record Dates: First submitted 2022-01-08; First posted 2022-02-03 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age-related macular degeneration; AMD; Medical Eye Trainer
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
People with the disease age-related macular degeneration (AMD) are treated with the Medical Eye Trainer (MET) system to improve their vision. The training is carried out over 2 months.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is a widespread eye disease worldwide. According to the Gutenberg Health Study, about 7000000 people in Germany suffer from it. The numbers for Austria are to be assumed with 700000 due to the smaller population. There are two different forms of AMD, the wet form with 15% and the dry form with 85%. Both types have a high risk of rapid development of significant visual impairment. For the dry form of the disease there are currently only a few therapeutic options. The main one is the nutritional supplement therapy. This treatment can only reduce the progression of deterioration in 10% of affected individuals, but there is a significant side effect profile. Thus, the question arose for completely different treatment approaches. For this reason, the Medical Eye Trainer (MET) was developed. This is a training device which can easily be used in self application. The purpose of this new therapy is not to try to cure AMD. Instead, the eye and brain are trained to better cope with the disease. In a first study on 17 eyes, 11 cases even showed an improvement of the visual performance, the remaining 6 cases showed a stable situation. In no case did a deterioration occur. Thus, for the first time, it was possible not only to slow down this disease, but even to achieve an improvement. In a second study with a planned number of 150 persons, this positive effect will be further investigated. A calculation with G*Power, based on the results of the first study, results in an optimal number of 150 examinations.

The participants will be examined in the hospital Ried im Innkreis and treated by MET. No additional measures are required for the study besides the usual eye examinations in AMD.

The study is open to individuals with dry AMD, regardless of age. Exclusion criteria are wet AMD, epilepsy and double vision. Other eye diseases are not a problem.

The diagnosis is additionally confirmed by an examination of the ocular fundus with an Optical Coherence Tomography (OCT). As an essential factor of the severity of the disease, the visual performance for distance (5-6m) and for near (40cm) is determined.

Participants need a mobile electronic device with the operating system Apple IOS® or Android®. The MET training system in the form of software will be provided for the duration of the study. The therapy is performed daily by the patient him/herself and lasts 90 seconds per eye. A success control is planned after two months. The above mentioned examinations will be repeated.

The MET has a CE-approval in the sense of MPG class 1. This study will be performed according to the Helsinki criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age-related macular degeneration

Exclusion Criteria:

* Epilepsy
* Double vision

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All persons with dry AMD who have no risk of reacting to the intense visual stimulus with a seizure. Existing double images are intensified by the increased visual acuity. All other affected persons can participate in the training.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in visual acuity | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- BHS Ried, Ried im Innkreis, Upperaustria, Austria

IPD SHARING:
Plan to Share IPD: No
Based on the European Data Protection Regulation, no data transfer is allowed.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT05222997/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT05222997/ICF_001.pdf